CLINICAL TRIAL: NCT04434300
Title: Comparison of the Pharmacokinetic and the Safety of Daptomycin Administered Subcutaneously Compared to the Intravenous Route : a Cross-over Study
Brief Title: Subcutaneous Daptomycin in Healthy Volunteers (DAPTOSC)
Acronym: DAPTOSC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-004884-32
Record Dates: First submitted 2020-04-29; First posted 2020-06-16 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2021-07

CONDITIONS: Antibiotics; Subcutaneous Injection; Daptomycin
MeSH Terms: interventions — Daptomycin

STUDY DESIGN:
Who Masked: Participant
Masking Description: Subcutaneous administration of daptomycin and placebo will be done blind to the participant. Given the yellow coloration of daptomycin, a masking of the pockets of daptomycin and NaCl will be carried out with a pocket cover and an opaque tube will be used for the administration
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapto SC-IV (Other): First stage :
  * Subcutaneous injection of daptomycin 10mg/kg
  * Subcutaneous injection of placebo (physiological serum)
  Second stage :
  - Intravenous injection of daptomycin 10mg/kg
  Interventions: Drug: Daptomycin
- Dapto IV-SC (Other): First stage :
  - Intravenous injection of daptomycin 10mg/kg
  Second stage :
  * Subcutaneous injection of daptomycin 10mg/kg
  * Subcutaneous injection of placebo (physiological serum)
  Interventions: Drug: Daptomycin

INTERVENTIONS:
Drug: Daptomycin — Compare the pharmacokinetic of subcutaneous (SC) and intravenous (IV) routes in the same patient.
  Arms: Dapto SC-IV
Drug: Daptomycin — Compare the pharmacokinetic of subcutaneous (SC) and intravenous (IV) routes in the same patient.
  Arms: Dapto IV-SC

SUMMARY:
Background:

Multidrug-resistant bacteria are a major public health problem worldwide, notably due to excess mortality and an increase in the length of hospital stay. Antibiotics that can be used to treat these infections are limited. Daptomycin is one of the most widely used antibiotics for the treatment of infections with gram-positive bacteria, such as methicillin-resistant Staphylococcus aureus (MRSA). However, it is only administered intravenously (IV). It is therefore interesting to find new routes of administration in order to widen the possibilities of using daptomycin, especially in people who have difficulties with the venous approach.

Methods/design:

In a randomized, single blinded, crossover, noninferiority study in the CHU of Caen, the investigators aim to demonstrate the pharmacokinetic bioequivalence between the subcutaneous and the intravenous route of daptomycin in healthy volunteers. They will conclude the bioequivalence if the confidence interval of the area under the curve obtained is entirely within the interval [80% - 125%].

Discussion:

This clinical trial could, if bioequivalence is demonstrated, lead to the completion of a clinical trial in infected patients in order to assess the efficacy and safety of daptomycin by the subcutaneous route.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer from 18 to 65 years old
* Subject determined in good health by a doctor
* Signature of free and informed consent
* Affiliated to the French healthcare insurance
* Fluent in French

Exclusion Criteria:

* Active bacterial or viral infection
* Immunocompromised
* Body mass index <20 or> 30 kg / m2
* Kidney failure with glomerular filtration rate <90ml / min / m2 calculated according to the CKD-EPI method
* Known or suspected liver disease
* Pregnant or lactating woman
* Guardianship or curators
* Any situation that could interfere with the self / hetero assessment of pain (dementia, psychiatric disorders, for example)
* Concomitant intake of myotoxic drugs (statins, fibrates, ciclosporin, for example)
* Allergy or known side effects to daptomycin
* Dermatological pathologies which may interfere with the subcutaneous injection (eczema, psoriasis, etc.)
* Localized tattoo or piercing on the abdomen which may interfere with the subcutaneous injection or the evaluation of possible local effects of the injection
* Parenteral exposure to daptomycin in the previous 30 days
* The inclusion of the subject in another interventional research protocol (during the present study and in the 3 months before inclusion).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
daptomycin dosage after intravenous route | before injection
  measurement of daptomycin blood concentration after intravenous route
daptomycin dosage after intravenous route | 30 minutes after injection
  measurement of daptomycin blood concentration after intravenous route
daptomycin dosage after intravenous route | 1 hours after injection
  measurement of daptomycin blood concentration after intravenous route
daptomycin dosage after intravenous route | 1,50 hours after injection
  measurement of daptomycin blood concentration after intravenous route
daptomycin dosage after intravenous route | 2 hours after injection
  measurement of daptomycin blood concentration after intravenous route
daptomycin dosage after intravenous route | 3 hours after injection
  measurement of daptomycin blood concentration after intravenous route
daptomycin dosage after intravenous route | 4 hours after injection
  measurement of daptomycin blood concentration after intravenous route
daptomycin dosage after intravenous route | 8 hours after injection
  measurement of daptomycin blood concentration after intravenous route
daptomycin dosage after intravenous route | 10 hours after injection
  measurement of daptomycin blood concentration after intravenous route
daptomycin dosage after intravenous route | 24 hours after injection
  measurement of daptomycin blood concentration after intravenous route
daptomycin dosage after subcutaneous route | before injection
  measurement of daptomycin blood concentration after subcutaneous route
daptomycin dosage after subcutaneous route | 30 minutes after injection
  measurement of daptomycin blood concentration after subcutaneous route
daptomycin dosage after subcutaneous route | 1 hours after injection
  measurement of daptomycin blood concentration after subcutaneous route
daptomycin dosage after subcutaneous route | 1.50 hours after injection
  measurement of daptomycin blood concentration after subcutaneous route
daptomycin dosage after subcutaneous route | 2 hours after injection
  measurement of daptomycin blood concentration after subcutaneous route
daptomycin dosage after subcutaneous route | 3 hours after injection
  measurement of daptomycin blood concentration after subcutaneous route
daptomycin dosage after subcutaneous route | 4 hours after injection
  measurement of daptomycin blood concentration after subcutaneous route
daptomycin dosage after subcutaneous route | 8 hours after injection
  measurement of daptomycin blood concentration after subcutaneous route
daptomycin dosage after subcutaneous route | 10 hours after injection
  measurement of daptomycin blood concentration after subcutaneous route
daptomycin dosage after subcutaneous route | 24 hours after injection
  measurement of daptomycin blood concentration after subcutaneous route

SECONDARY OUTCOMES:
Local adverse events | within the first 24hours after injection
  Occurrence of local adverse events (pain, erythema, edema, necrosis)
Local adverse events | 3 days after the infusion
  Occurrence of local adverse events (pain, erythema, edema, necrosis)
Local adverse events | 7 days after the infusion
  Occurrence of local adverse events (pain, erythema, edema, necrosis)
Systemic adverse events | within the first 24hours after injection
  Occurrence of systemic adverse events
Systemic adverse events | 3 days after the infusion
  Occurrence of systemic adverse events
Systemic adverse events | 7 days after the infusion
  Occurrence of systemic adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Caen, Caen, Normandy, France

REFERENCES:
- [Derived] Maurille C, Baldolli A, Creveuil C, Parienti JJ, Michon J, Peyro-Saint-Paul L, Brucato S, Dargere S, Comets E, Verdier MC, Verdon R. Pharmacokinetics and safety of daptomycin administered subcutaneously in healthy volunteers: a single-blinded randomized crossover trial. J Antimicrob Chemother. 2024 Nov 4;79(11):3016-3022. doi: 10.1093/jac/dkae324. PMID 39271104